CLINICAL TRIAL: NCT05664854
Title: Electrical Impedance Tomography Imaging of Functional Anatomy and Selective Stimulation of Fascicles Within the Vagus Nerve
Brief Title: Electrical Impedance Tomography & Selective Stimulation of Vagus Nerve
Acronym: EITsVNS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kirill Aristovich, Associate Professor, University College, London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 275276; 3OT2OD026545 (NIH); 147583 (Other: UCL Sponsor Reference Number - EDGE); 22/LO/0463 (Other: REC Reference); Z6364106/2022/03/39 (Other: Social Research Number)
Record Dates: First submitted 2022-12-02; First posted 2022-12-27 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Vagus Nerve Diseases; Epilepsy; Vagus Nerve Autonomic Disorder
Keywords: Electrical Impedance Tomography; Selective Vagus Nerve Stimulation; Vagus Nerve; Electrophysiology; Vagus Nerve Stimulation
MeSH Terms: conditions — Vagus Nerve Diseases; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sVNS and EIT of cervical vagus nerve (Experimental): Selective vagus nerve stimulation (sVNS) with a spatially selective vagal nerve cuff with physiological readouts such as electrocardiogram (ECG), heart rate, end-tidal carbon dioxide (EtCO2), respiratory rate, laryngeal electromyogram (EMG), etc., and electrical impedance tomography (EIT) recordings of the nerve.
  Interventions: Device: Nerve cuff electrodes for spatially selective vagus nerve stimulation and electrical impedance tomography

INTERVENTIONS:
Device: Nerve cuff electrodes for spatially selective vagus nerve stimulation and electrical impedance tomography — Vagus nerve electrode cuffs will be placed on the exposed human vagus nerve during routine vagal nerve stimulator implantation surgery. These cuffs will then be used for spatially selective vagus nerve stimulation, with physiological readout, and electrical impedance tomography for the functional imaging of organ-specific regions in the nerve at cervical level.

SUMMARY:
Electroceuticals is a new field in which the goal is to treat a wide variety of medical diseases with electrical stimulation of autonomic nerves. A prime target for intervention is the cervical vagus nerve as it is easily surgically accessible and supplies many organs in the neck, thorax and abdomen. It would be desirable to stimulate selectively in order to avoid the off-target effects that currently occur. This has not been tried in the past, both because of limitations in available technology but also because, surprisingly, the fascicular organisation of the cervical vagus nerve is almost completely unknown. The aim of this research is to investigate the functional anatomy of fascicles in the cervical vagus nerve of humans. This will include defining innervation to the heart, lungs and recurrent laryngeal and, if possible, the oesophagus, stomach, pancreas, liver and gastrointestinal tract. It will be achieved by defining fascicle somatotopic functional anatomy with spatially-selective vagus nerve stimulation (sVNS) and the new method of fast neural imaging with Electrical Impedance Tomography (EIT). EIT is a novel imaging method in which reconstructed tomographic images of resistance changes related to the opening of ion channels over milliseconds can be produced using rings or arrays of external electrodes. In humans, using a nonpenetrating nerve cuff with sVNS or fast neural EIT, this will be performed for 30 minutes transiently during an operation to insert a vagal nerve stimulator for treatment of epilepsy and deliver images in response to activity such as respiration or the electrocardiogram (ECG).

DETAILED DESCRIPTION:
Electroceuticals is a relatively new field in which the goal is to treat a wide variety of medical diseases with electrical stimulation of autonomic nerves. A prime target for intervention is the cervical vagus nerve as it is easily surgically accessible and supplies many organs in the neck, thorax and abdomen. It would be desirable to stimulate selectively in order to avoid the off-target effects that currently occur. Until recently, this has not been tried in the past, both because of limitations in available technology but also because, surprisingly, the fascicular organisation of the cervical vagus nerve is almost completely unknown; work has recently been performed in animal models. The aim of this research is to investigate the functional anatomy of fascicles (groups of nerve fibres) in the cervical vagus nerve of humans. This will include defining innervation to the heart, lungs and recurrent laryngeal and, if possible, the oesophagus, stomach, pancreas, liver and gastrointestinal tract. After the specific locations of above groups are identified, it will be possible to direct the stimulation so that only specific organs are affected by the vagus nerve stimulation. In particular, it may be possible to achieve a therapeutic seizure-suppressive effect in Epilepsy with better efficacy, and, at the same time, avoid all side effects normally present because all of the organ functions are altered when the entire nerve gets stimulated.

Our group has pioneered the use of a multi-purpose nerve cuff for imaging activity within nerves with Electrical Impedance Tomography (EIT) and with the ability of spatially-selective neuromodulation. It has been optimised and validated for use in vivo in animal models.

Vagus nerve stimulation (VNS) is currently perform in humans for the treatment of drug-resistant epilepsy and depression. However, VNS as a therapeutic intervention can be expanded to a vast range of therapeutic applications. Ongoing studies and preclinical research indicate promising results in treating cardiovascular disorders and heart failure, lung injury, asthma, sepsis, rheumatoid arthritis, diabetes, obesity, pain management and targeting the anti-inflammatory pathway in general. In addition, selective neuromodulation could be used as a therapeutic approach for the treatment of acute respiratory distress syndrome, predominant currently during the Covid-19 pandemic, which requires the activation of some pathways (cholinergic anti-inflammatory pathway) and not others (pulmonary function) to effectively improve outcomes.

Even with the vast potential of VNS in treating a variety of diseases, limitations still exist. Without the knowledge of the neuroanatomy of the target nerve, side effects prevail and reduce the efficacy of treatment. A large proportion of side-effects frequently experienced, including cough, dyspnoea and hoarseness, can be attributed to activation of the recurrent laryngeal nerve fibres in the vagus nerve. Avoidance of vagal outflow to the larynx alone could greatly improve VNS and reduce the side effects so often observed. However, knowledge of the innervation from all regions within the cervical vagus nerve could further improve targeted stimulation and therapeutic efficacy; avoiding any unwanted responses in non-targeted organs such as shortness of breath and bradycardia and could reduce the risk of further, long-term side effects, such as developing hyperglycaemia when stimulating for epilepsy.

EIT and selective stimulation of the human vagus nerve holds promise to provide information of the fascicular organisation of the nerve which would allow for targeted neuromodulation during the treatment of epilepsy, depression and other disorders without indiscriminate vagal outflow thereby avoiding off-target effects currently experienced. The efficacy and therapeutic outcomes of VNS will be improved. It requires interdisciplinary collaboration from biomedical scientists, electronic engineers and mathematicians, and holds great interest for those interested in interdisciplinary work in these fields.

During routine vagal nerve stimulator implantation surgery, the operating surgeon will place a temporary electrode cuff for the purpose of this study only, after gaining access to the vagus nerve. This cuff will be removed during the same surgery after the protocol has been completed, and the surgery completed as usual. This cuff is designed for single use, made of sterilised platinum and medical-grade silicone - a layer of platinum containing traces and electrodes arranged in rings is confined between two layers of medical-grade silicone. To ensure the cuff is in contact with the nerve, a medical-grade silicone support, in the form of a tube with an opening, or biocompatible clamps attached to the opening ends of the cuff will be used at the discretion of the surgeon. One end of the cuff has a connector leading to an electronic device that is used for the stimulations and recordings. Whilst the patient is still under for their routine implantation surgery, both selective stimulation and EIT recordings (imaging) will take place. An electrical current will be driven between a pair of electrodes present on the cuff, and the process will be repeated for different pairs while recording physiological parameters (ECG (recording of the heart activity), respiration, electrogastrogram) to look for physiological changes. Parameters, such as current, pulse width and frequency, will be adjusted to elicit responses in the nerve by different nerve fibre types. Stimulation will be performed for approximately up to 28 minutes (10 to 30 seconds per pair with waiting time in between to return to baseline). This may be repeated with different stimulation parameters. Subsequently, nerve imaging (EIT) will be performed in a similar way with current injected through various electrode pairs; however, this time other electrodes on the cuff will be used to record electrical properties, specifically impedance, from the nerve. This will take place for approximately 28 minutes as well. The cuff will be removed by the surgeon at the end of the protocol and the surgery will be completed as usual for the standard implantation surgery. This will complete the involvement of the patient in this study. All measurements and recordings will be analysed at a later stage by the researchers in their lab and office, to get information about selective vagus nerve stimulation and form images of the activity within the nerve and the level of cuff implantation.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Written informed consent by patient or proxy
* Clinical diagnosis of disorder affected directly or indirectly or will possibly respond to vagus nerve stimulation

Exclusion Criteria:

* Aged 17 and below
* Unfortunately, it is unlikely that interpreters of all languages will be available in the unit so persons who cannot understand verbal explanation in English and for whom we could not find a suitable consultee would have to be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome - Map of organ-specific functional activity in the cervical vagus nerve | Within the first 3 years
  The cross-sectional map of organ-specific fascicles within the cervical vagus, indicating the location of pulmonary, cardiac, and recurrent laryngeal fascicles. The response in the appropriate organ(s) along with the imaging of the fascicles within the cervical vagus nerve and the degree of accordance of this with the fascicular map will be the primary outcomes.

SECONDARY OUTCOMES:
Secondary Outcome - Optimised neurostimulation parameters | Within the first 4 years
  Achieved parameters of the neurostimulation such that measured biomarker effect for seizure suppression matches or exceeds that of a whole-nerve stimulation with conventional device, while side effects (heart rate change, pressure, respiratory reflexes, and laryngeal activity) are significantly decreased.
  The performance of selective stim VS existing technique is assessed with binary metric: success/no success. The success criteria is: The therapeutic biomarker is not significantly different from the existing technique, while there is a significant reduction in one of the biomarkers indicating the side effects. The exact therapeutic biomarker will be identified during execution of the first objective. The biomarkers indicating side effects: significant bradycardia, apnoea, laryngeal contraction, gastric motility. The effect is calculated as a % change of the measured physiological parameter during stimulation with respect to the baseline (no stimulation).

CONTACTS AND LOCATIONS:
Overall Officials: Kirill Aristovich, Principal Investigator — University College, London
Locations (1):
- National Hospital of Neurology and Neurosurgery, London, Greater London, United Kingdom